CLINICAL TRIAL: NCT00971568
Title: Urinary Biomarkers Characteristic to Interstitial Cystitis- Proteomic Analysis of Urine
Brief Title: Urinary Biomarkers Characteristic to Interstitial Cystitis
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-163
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Interstitial Cystitis
Keywords: Interstitial cystitis; Painful bladder syndrome
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Urine sample: To prepare for SELDI-TOF we will use 15 samples. Each sample (25ul) will be analyzed with the Luminex 100 IS (MiraiBio, South San Francisco, CA) using a LINCOplex cytokine/che-

SUMMARY:
This is a retrospective study of urine samples stored in the Beaumont BioBank for future research. The urine samples will be drawn from the urine back with patients previously diagnosed with severe interstitial cystitis (IC), mild IC and no IC.

Interstitial Cystitis (IC) also known as Painful Bladder Syndrome (PBS) is a chronic inflammatory disease. It has an unknown etiology, symptoms which present to varying degrees, as well as an uncertain natural history. Diagnosis of IC is based on symptoms after excluding more common and dangerous pathologies.

DETAILED DESCRIPTION:
Extensive research has been done to understand the multifactorial etiology as well as to help diagnose IC. Infectious, autoimmune and anatomic causes have been looked at with few usable results. Inflammatory cells and markers have been more productive. Recently we have shown in the rat model, that chemically induced inflammation, yields temporal increases in measurable cytokines and chemokines in the urine. Moreover, this was done by Multiplex analysis, using a multiple antigen bead assay (Luminex).

Cytokines and chemokines, part of an organisms proteome, allow for looking at the function of a cell or organ at the time of the collection United States: Institutional Review Board. Urine is obtained non-invasively and yields significant information about urinary tract organs. The ability to find a biomarker or pattern of biomarker in the urine, diagnostic to a disease, offers significant advantages over serum or tissue diagnosis.

We hope to identify patterns of inflammatory markers using proteomic analysis using the previously mentioned multiple antigen cassettes (Luminex) as well as identify possible new biomarkers using a Protein Chip SELDI--TOF (surface enhanced laser desorption ionisation-time of flight) mass spectrometer. The detection of patterns or new biomarkers has promise to help with diagnosis, treatment, and ultimately revealing the etiology and course of IC.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have previously been contacted and consented to place a sample within the biobank. We will select five representative patients from the severe IC diagnosis, mild IC diagnosis, and no IC diagnosis, and we will match these patients as best as possible within the limited biobank samples.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will be examining urine already collected and in the Beaumont Biobank. The urine to be examined is from patients with known severe Interstitial Cystitis (IC), mild IC or known to not have the disease.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Using a ProteinChip SELDI--TOF (surface enhanced laser desorption ionisation-time of flight) mass spectrometer, we will analyze previously collected urine samples from matched patients with severe IC, mild IC and controls without disease. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chancellor, MD, Principal Investigator — Beaumont Hospitals
Locations (1):
- Beaumont Hospitals-Royal Oak, Royal Oak, Michigan, United States